CLINICAL TRIAL: NCT03500913
Title: Adipose Tissue and Serum Inflammation in Growth Hormone (GH) Deficiency
Brief Title: Adipose Tissue and Serum Inflammation in GH Deficiency
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Pamela U. Freda, Professor of Medicine, Columbia University
Other Study IDs: AAAP3950; 1R01DK110771-01A1 (NIH)
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Growth Hormone Deficiency
Keywords: Growth Hormone Deficiency; Adipose Tissue; Inflammation
MeSH Terms: conditions — Dwarfism, Pituitary; Inflammation | interventions — Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Peripheral venous blood
  2. Subcutaneous adipose tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adults with growth hormone deficiency: Subjects who present to the neuroendocrine unit at Columbia University Irving Medical Center (CUIMC) for therapy of GH deficiency or who are followed in the unit and have active GH deficiency and are planning to initiate a therapy.
  Interventions: Drug: Growth Hormone
- Control group: Healthy subjects matched to the GH deficiency subjects for age (+/- 5 years), gender and total fat mass (+/- 4%).

INTERVENTIONS:
Drug: Growth Hormone — Patients will receive growth hormone replacement therapy as per standard clinical care during this study.
  Other Names: GH
  Groups: Adults with growth hormone deficiency

SUMMARY:
This study will examine adipose tissue inflammation and adipokine expression and serum markers of inflammation and adipokine levels in patients with growth hormone (GH) deficiency before and after treatment.

DETAILED DESCRIPTION:
The GH axis has important influences on adipose tissue. Preliminary data from the investigators' study in acromegaly, a state of GH excess, suggests that GH reduces adipose tissue (AT) mass and serum inflammation. However, GH seems to reduce macrophage markers in adipose tissue yet increase adipocyte inflammation. This novel dissociation of macrophage and adipocyte inflammation is hypothesized to be due to GH. In order to examine this hypothesis further this study will examine adipose tissue and serum inflammation in patients with GH deficiency before and after GH therapy. The investigators will obtain subcutaneous adipose tissue by biopsy in patients with active GH deficiency planning to undergo therapy for GH deficiency. Concurrently serum samples will be taken for analysis of levels of inflammatory markers and adipokines. After treatment for 12 months with a normal levels of Insulin-like growth factor 1 (IGF-1), a marker of GH deficiency, patients will have a repeat adipose tissue biopsy. Adipose tissue parameters will be analyzed in each specimen and then compared to each patient over time as well as to body mass index (BMI)-matched control subjects.

ELIGIBILITY:
Inclusion criteria:

1. Males or females age ≥18 years with diagnosis of GH deficiency that is Adult Onset, either alone or associated with multiple pituitary hormone deficiencies and due to pituitary disease,hypothalamic disease, surgery, radiation therapy or Childhood Onset due to congenital, genetic, acquired, or idiopathic causes.
2. Diagnosis of GH deficiency defined by: insulin tolerance test or glucagon test: peak growth hormone response < 3 ng/ml or 3 or more pituitary hormone deficiencies and IGF-1 standard deviation score < -2.0
3. No history of diabetes mellitus and fasting blood sugar at screening visit ≤ 120 mg/dl.
4. If patients have undergone surgical resection of a pituitary adenoma, a minimum of 12 months must have elapsed post surgery prior to enrollment and tumor will be demonstrated to be unchanged for 12 months or longer since surgery.
5. May have a history of radiotherapy, but they must have completed their course of radiotherapy more than 3 months prior to study screening.
6. If prior GH therapy must have not received prior growth hormone replacement therapy in 310 the 6 months prior to screening.
7. Stable pituitary hormone supplements (x 3 months) prior to baseline visit and normal levels of free thyroxine, testosterone in males and normal adrenal function if not on replacement therapy.
8. If female, a. Not pregnant (as evidenced by a negative serum pregnancy test) or lactating and b. If of childbearing potential, agrees to use a medically acceptable form of contraception (such as oral, implantable, or barrier contraception) from the time of screening, for the duration of the study, and for at least one month after study discontinuation or completion. Childbearing potential is defined as women who are not surgically sterile or not at least one year postmenopausal.
9. Sign and date an informed consent document indicating that the subject (or legally acceptable representative) has been informed of and agrees to all pertinent aspects of the trial.

Exclusion Criteria:

1. Have other conditions that may result in abnormal GH and/or IGF-I concentrations (e.g., severe hepatic disease, severe renal disease, malnutrition, treatment with levodopa).
2. Alanine aminotransferase (ALT) or aspartate transaminase (AST) ≥ 2 x upper limit of normal or clinically significant hepatic disease or renal impairment defined as creatinine > 1.5x upper normal.
3. Have a pituitary adenoma with a distance to the optic chiasm of 5 mm or less, confirmed by a recent MRI scan (within two months prior to the screening visit).
4. Pituitary tumor growth within the 12 months prior to study entry.
5. GH therapy within 6 months of screening.
6. Diabetes mellitus.
7. History of acromegaly.
8. History of active Cushing's disease within 24 months of screening
9. Visual field defects or other neurological symptoms due to current tumor mass compression.
10. Have known or suspected drug or alcohol abuse.
11. Have received an investigational medication within four weeks prior to Screening or is scheduled to receive any investigational medication during the study.
12. Do not have the ability to fully comprehend the nature of the study, to follow instructions, cooperate with study procedures, and/or are unable to adhere to the visit scheduled outlined in the protocol.
13. Have other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
14. History of a malignancy other than squamous or basal cell skin carcinoma that has been excised or intracranial malignant tumors or leukemia within 5 years of screening.
15. Patients who have a known hypersensitivity to growth hormone therapy
16. Use of weight 349 loss medications
17. Females who plan to change estrogen therapy during the trial
18. Patients who have received supraphysiologic doses of glucocorticoids within the past 6 months (except for peri-operative (< 3 days duration) of dexamethasone), or who are currently receiving any chemotherapeutic agents.
19. Patients who have received other investigational drugs administered or received within 30 days of study entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential subjects include all those who present to our Neuroendocrine Unit for therapy of GH deficiency or who are followed in our unit and have GH deficiency and are planning to initiate a therapy. Subjects will be those with central adiposity. We expect are study group to be approximately half women and reflect the ethnic mix of our study populations of our other pituitary tumor studies, which is primarily drawn from the New York Metropolitan area.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2019-05-19 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Visceral Adipose Tissue (VAT) mass | Baseline to 12 months of GH therapy
  Visceral adipose tissue mass as measured by tota body magnetic resonance imaging

SECONDARY OUTCOMES:
Intra-hepatic lipid level | Baseline to 12 months of GH therapy
  Intra-hepatic lipid level measured by magnetic resonance imaging of liver
Skeletal Muscle Mass | Baseline to 12 months of GH therapy
  Skeletal muscle mass measured by total body magnetic resonance imaging
Total body fat | Baseline to 12 months of GH therapy
  Total body fat as measured by dual x-ray absorptiometry
Resting metabolic rate | Baseline to 12 months of GH therapy
  Resting metabolic rate
Relative gene expression of CD68 gene | Baseline to 12 months of GH therapy
  Relative gene expression values of Cluster of Differentiation 68 (CD68) gene expression in adipose tissue
Relative gene expression values of MCP1 gene | Baseline to 12 months of GH therapy
  Relative gene expression values of monocyte chemoattractant protein-1 (MCP-1) gene in adipose tissue
Relative gene expression IL6 gene | Baseline to after 12 months of treatment for GH deficiency
  Relative gene expression Interleukin 6 (IL6) gene in adipose tissue
Relative gene expression values of CD11c gene | Baseline to 12 months of GH therapy
  Relative gene expression values of CD11c gene in adipose tissue
interleukin 6 (IL-6) level | Baseline to 12 months of GH therapy
  Plasma level of interleukin 6 (IL-6)
TNFα level | Baseline to 12 months of GH therapy
  Plasma level of tumor necrosis factor alpha (TNFα)
CRP level | Baseline to 12 months of GH therapy
  Plasma level of C-reactive protein (CRP)
homocysteine level | Baseline to 12 months of GH therapy
  Plasma level of homocysteine

CONTACTS AND LOCATIONS:
Overall Officials: Pamela U. Freda, MD, Principal Investigator — Columbia University
Locations (1):
- Neuroendocrine Unit and Pituitary Center, Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided